CLINICAL TRIAL: NCT03770312
Title: Low- and Moderate-intensity Statin and Clinical Outcome of Primary Prevention in Individuals Aged >70 Years: the SCOPE-70 RCT Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2019-1219
Record Dates: First submitted 2018-12-04; First posted 2018-12-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Elderly Individuals With High LDL-cholesterol or Risk of Cardiovascular Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low intensity statin group (Active Comparator): Taking low intensity statin
  Interventions: Drug: Low intensity statin
- Moderate intensity statin group (Active Comparator): Taking moderate intensity statin
  Interventions: Drug: Moderate intensity statin

INTERVENTIONS:
Drug: Low intensity statin — Use of low intensity statin for primary prevention of cardiovascular disease.
  Arms: Low intensity statin group
Drug: Moderate intensity statin — Use of moderate intensity statin for primary prevention of cardiovascular disease.
  Arms: Moderate intensity statin group

SUMMARY:
One of the most effective drug in the primary prevention of cardiovascular disease is statins. The protective effects of statin on developement of cardiovascular disease has been demonstrated in elderly individuals. Since side effects of statin are more common in elderly individuals than in younger individuals, clinical guidelines recommend that use of low intensity statin is considered in elderly individuals. However, there are few randomized clinical trials evaluating the safety and efficacy of different intensity statins in elderly individuals.

This is a multicenter, prospective, randomized clinical trial to compare efficacy and safety between low and high intensity statin for primary prevention of cardiovacsular disease in elderly individuals.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized clinical trial evaluating the safety of low-intensity statins versus moderate-intensity statins in the primary prevention of cardiovascular disease in elderly patients aged 70 years or older without cardiovascular disease. The patient recruitment period is 2 years, with a 6-month follow-up period (a 4-year follow-up is optional).

Individuals deemed eligible through screening will be randomly assigned in a 1:1 ratio to either the rosuvastatin 2.5mg or rosuvastatin 10mg group. After randomization, subjects will visit at 3 and 6 months for scheduled blood tests, physical examinations, and questionnaires regarding muscle symptoms. After 6 months, subjects may optionally continue routine primary cardiovascular disease prevention care for a total of 4 years of follow-up.

ELIGIBILITY:
"Inclusion criteria

1. Adults aged 70 years or older as of the date of written consent, meeting one of the criteria in items 2-5)
2. Patients with no prior statin use or who have discontinued statin therapy for at least 4 weeks, with no cardiovascular risk factors* and LDL-cholesterol levels of 160-189 mg/dL
3. Patients with no prior statin use or who have discontinued statins for at least 4 weeks, with one or more cardiovascular disease risk factors* and LDL-cholesterol levels of 80-189 mg/dL
4. For patients currently taking statins, with 0 cardiovascular disease risk factors* and LDL-cholesterol levels of 95-114 mg/dL
5. For patients currently taking statins, with 1 or more cardiovascular disease risk factors* and LDL-cholesterol levels of 50-114 mg/dL

   * Cardiovascular Disease Risk Factors

     * Male
     * Family history of early cardiovascular disease: myocardial infarction, angina, peripheral vascular disease, ischemic stroke; men <55 years, women <65 years
     * Diabetes: One or more of the following five criteria: HbA1c ≥6.5%, fasting blood glucose ≥126 mg/dL, postprandial 2-hour blood glucose ≥200 mg/dL, random blood glucose ≥200 mg/dL with typical symptoms like polyuria, or the use of antidiabetic medication
     * Hypertension: Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, or use of antihypertensive medication
     * Current smoker
     * HDL-cholesterol <40 mg/dL

Exclusion criteria (any):

1. Individuals who have been diagnosed with cancer within the last 5 years.
2. Individuals who have high level of serum ALT (>2 upper normal limit).
3. Individuals who have serum creatinine ≥2 mg/dL.
4. Individuals who have been diagnosed with cardiovascular disease (>50% stenosis of coronary artery on imaging study, percutaneous transluminal coronary angioplasty, coronary artery bypass graft, or myocardial infarction).
5. Individuals who have been diagnosed with peripheral artery disease (>50% stenosis of peripheral artery on imaging study, or ankle brachial index <0.9 or ≥1.3).
6. Individuals who have been diagnosed with uncontrolled hyperthyrodism or hypothyroidism.
7. Individuals who are taking drug that can interact with statin.
8. Individuals who have physical disability to live daily life.
9. Individuals with genetic disorders such as galactose intolerance (including preparations containing lactose)"

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 724 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Statin associated muscle symptoms (SAMS) -If all of the following occur, it is defined as SAMS. | 3 months
  1. They report new or increased myalgia, cramps, or muscle aching, unassociated with recent exercise.
  2. These symptoms have persisted for at least 2 weeks.
  3. The symptoms resolve within 2 weeks of stopping the study drug.
  4. The symptoms reoccur within 4 weeks of restarting the medication.
Statin associated muscle symptoms (SAMS) -If all of the following occur, it is defined as SAMS. | 6 months
  1. They report new or increased myalgia, cramps, or muscle aching, unassociated with recent exercise.
  2. These symptoms have persisted for at least 2 weeks.
  3. The symptoms resolve within 2 weeks of stopping the study drug.
  4. The symptoms reoccur within 4 weeks of restarting the medication.
Statin associated muscle symptoms (SAMS) - Statin associated muscle symptoms are judged using the Short-Form Brief Pain Inventory (BPI-SF). | 3 months
Statin associated muscle symptoms (SAMS) - Statin associated muscle symptoms are judged using the Short-Form Brief Pain Inventory (BPI-SF). | 6 months
Statin associated muscle symptoms (SAMS) - Statin associated muscle symptoms are judged using the Short-Form McGill Pain Questionnaire (SF-MPQ) | 3 months
Statin associated muscle symptoms (SAMS) - Statin associated muscle symptoms are judged using the Short-Form McGill Pain Questionnaire (SF-MPQ) | 6 months

SECONDARY OUTCOMES:
Clinical outcomes | 4 years for MACE. 6 months for all adverse events.
  Major adverse cardiovascular events, defined as the composite endpoint comprised of cardiovascular death, nonfatal MI, nonfatal ischemic stroke, TIA, coronary revascularization (PCI or CABG), or hospitalization for unstable angina during extended follow-up up to 48 months.
  All adverse events during 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Cardiovascular Center, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No